CLINICAL TRIAL: NCT01081340
Title: Building Social Networks to Enhance Postpartum Weight Loss and Appropriate Infant Feeding Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00034677
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: gestational weight gain; postpartum weight loss; breastfeeding; overfeeding
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Breast Feeding | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social network building intervention (Experimental): Healthy lifestyle intervention focused on building reciprocal social ties between the intervention group members
  Interventions: Behavioral: Social network building intervention
- Home visit (Active Comparator): Home visits focused on preventable infant injuries
  Interventions: Behavioral: Home visit

INTERVENTIONS:
Behavioral: Social network building intervention — Group support and health education sessions weekly during third trimester and once every two weeks until 6 months postpartum
  Arms: Social network building intervention
Behavioral: Home visit — Three home visits during third trimester and three during postpartum period until 6 months postpartum
  Arms: Home visit

SUMMARY:
The purpose of this study is to examine whether we can use social networks to spread health information and health behaviors that 1) support women in returning to their pre-pregnancy weight after delivery; and 2) promote healthy infant feeding practices.

DETAILED DESCRIPTION:
The long-term goal of this research is to prevent obesity-related adverse health outcomes for future generations by applying information emerging from social network studies to the development of new population-based behavioral interventions. There are a number of critical periods during fetal and infant development that appear to influence the later development of obesity. Interventions that prevent insult to these critical windows from occurring could improve children's life course trajectories. This project sets the groundwork for examining whether social networks could explicitly be utilized to prevent obesity from developing by transmitting health information and health behaviors that 1) prevent postpartum weight retention in first time mothers and 2) promote appropriate infant feeding practices. The secondary aim is to assess which individual-level network-related characteristics best predict postpartum body composition and infant feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Latina (self-defined, or born in Central or South America)
* Spanish-speaking and/or English-speaking,
* 18 years of age or older
* less than 24 weeks pregnant
* did or did not have a termination of a previous pregnancy before 20 weeks
* has not carried a pregnancy to term
* normal, overweight or obese (pre-pregnancy BMI >18.5 and <39)

Exclusion Criteria:

* non-Latina,
* non-Spanish-speaking or non-English speaking
* less than 18 years of age
* more than 24 weeks pregnant
* had a termination of a previous pregnancy after 20 weeks
* multiparous
* underweight (pre-pregnancy BMI < 18.5)
* morbidly obese (pre-pregnancy BMI ≥ 39)
* currently enrolled in another program that targets weight, physical activity, or nutrition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Weight (kg) | 6 times over 10 months
  gestational weight gain and postpartum weight loss

SECONDARY OUTCOMES:
Body composition | 3 times over 6 months
  BIA postpartum
Infant feeding practices | 3 times over 6 months
  duration of breastfeeding, use of supplemental fluids, overfeeding, timing of the introduction of solids
Social network structure | 6 times over 10 months
  number and type of relationships
Waist Circumference | 3 times over 6 months
Depression | 6 times over 10 months
Nutrition | 6 times over 10 months
  Fat/Fruit/Vegetable intake
Physical Activity | 6 times over 10 months
  self-report

CONTACTS AND LOCATIONS:
Overall Officials: Sabina B Gesell, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Coleman Regional Community Center - Parks & Rec Department, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No